CLINICAL TRIAL: NCT06216847
Title: Clinical Outcomes of Patients With Coronary Artery Disease Cohort Study
Brief Title: Clinical Outcomes of Patients With Coronary Artery Disease
Acronym: COCAD
Status: Recruiting | Type: Observational
Sponsor: Shenyang Northern Hospital (Other)
Responsible Party: Principal Investigator, Han Yaling, Prof., Shenyang Northern Hospital
Other Study IDs: COCAD V1.0
Record Dates: First submitted 2024-01-11; First posted 2024-01-22 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Coronary Heart Disease (CHD)
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Coronary heart disease (CHD) stands as a foremost contributor to global mortality, characterized by complex pathogenesis that renders conventional "one-size-fits-all" preventive strategies inefficient. Therefore, the investigators designed a prospective, multi-center cohort study among patients hospitalized due to either confirmed or suspected CHD, which aimed to establish a holographic data set for the diagnosis and treatment of CHD and explore the impact of critical therapeutic strategies in the real world on the clinical outcomes of CHD patients, providing evidence to optimize the management pathway.

DETAILED DESCRIPTION:
Coronary heart disease (CHD) stands as a foremost contributor to global mortality. Despite the increasing investment in the prevention of risk factors and the popularization of percutaneous coronary intervention (PCI), the age-standardized incidence and mortality of CHD continue to increase. CHD is characterized by complex pathogenesis, rendering conventional "one-size-fits-all" preventive strategies inefficient.

Currently, there is a need to address two critical challenges. The first centers on early detection, precise risk stratification, and personalized intervention strategies for high-risk CHD patients, with a focus on the exploration of inflammation-driven risks, lesion-based risk stratification, and tailored anti-thrombotic therapies. The second challenge lies in the transformation of clinical risk assessment and decision-making processes into a precise level through the utilization of big data mining techniques.

Therefore, the investigators designed a prospective, multi-center cohort study among patients hospitalized due to either confirmed or suspected CHD, which aimed to establish a holographic data set for the diagnosis and treatment of CHD and explore the impact of critical therapeutic strategies in the real world on the clinical outcomes of CHD patients, providing evidence to optimize the management pathway.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Hospitalization due to either confirmed or suspected CHD combined with one of the following features: previous PCI or CABG; previous myocardial infarction; previous coronary angiography revealing ≥ 50% stenosis in major coronary vessels; presentation with chest pain and pre-test probability of CHD > 65%; laboratory tests revealing objective evidence of myocardial ischemia; coronary CT angiography (CTA) showed ≥ 30% stenosis in major coronary vessels
* Subjects undergoing at least one coronary imaging and one functional examination. Imaging examinations include coronary CTA, intravascular ultrasound (IVUS), or optical coherence tomography (OCT). Functional examination include fraction flow reservation (FFR), CT-FFR or quantitative flow ratio (QFR).
* Written informed consent provided.

Exclusion Criteria:

* History of mental illness, drug or alcohol abuse, or being unable to cooperate with follow-up visits for any reason;
* Life expectancy <1 year
* Pregnant or plan to be pregnant within 1 year
* Subjects participating in any other clinical trial
* Other conditions deemed unsuitable for inclusion by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients hospitalized due to either confirmed or suspected CHD
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2024-02-21 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2030-10-31 (Estimated)

PRIMARY OUTCOMES:
Ischemic events | During 12-month follow up
  defined as the composite of cardiac death, myocardial infarction, or stroke

SECONDARY OUTCOMES:
Major adverse cardiovascular and cerebrovascular events (MACCE) | During 1/2/3/4/5-year follow up
  defined as a composite of all-cause death, myocardial infarction, ischemic stroke and target-vessel revascularization
Cardiac death | During 1/2/3/4/5-year follow up
Stent thrombosis | During 1/2/3/4/5-year follow up
Major bleeding events | During 1/2/3/4/5-year follow up
  defined as BARC types 3 or 5 bleeding events
Clinical relevant bleeding events | During 1/2/3/4/5-year follow up
  defined as BARC type 2-5 bleeding events

CONTACTS AND LOCATIONS:
Overall Officials: Yaling Han, MD, Principal Investigator — The General Hospital of Northern Theater Command
Locations (1):
- General Hospital of Northern Theater Command, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liu S, Li Y, Zeng X, Wang H, Yin P, Wang L, Liu Y, Liu J, Qi J, Ran S, Yang S, Zhou M. Burden of Cardiovascular Diseases in China, 1990-2016: Findings From the 2016 Global Burden of Disease Study. JAMA Cardiol. 2019 Apr 1;4(4):342-352. doi: 10.1001/jamacardio.2019.0295. PMID 30865215
- [Background] writing committee of the report on cardiovascular health and diseases in china. Report on Cardiovascular Health and Diseases in China 2021: An Updated Summary. Biomed Environ Sci. 2022 Jul 20;35(7):573-603. doi: 10.3967/bes2022.079. PMID 35945174
- [Background] Currie G, Delles C. Precision Medicine and Personalized Medicine in Cardiovascular Disease. Adv Exp Med Biol. 2018;1065:589-605. doi: 10.1007/978-3-319-77932-4_36. PMID 30051409
- [Background] Liberale L, Badimon L, Montecucco F, Luscher TF, Libby P, Camici GG. Inflammation, Aging, and Cardiovascular Disease: JACC Review Topic of the Week. J Am Coll Cardiol. 2022 Mar 1;79(8):837-847. doi: 10.1016/j.jacc.2021.12.017. PMID 35210039
- [Background] Marnell CS, Bick A, Natarajan P. Clonal hematopoiesis of indeterminate potential (CHIP): Linking somatic mutations, hematopoiesis, chronic inflammation and cardiovascular disease. J Mol Cell Cardiol. 2021 Dec;161:98-105. doi: 10.1016/j.yjmcc.2021.07.004. Epub 2021 Jul 21. PMID 34298011
- [Background] Ridker PM, Everett BM, Thuren T, MacFadyen JG, Chang WH, Ballantyne C, Fonseca F, Nicolau J, Koenig W, Anker SD, Kastelein JJP, Cornel JH, Pais P, Pella D, Genest J, Cifkova R, Lorenzatti A, Forster T, Kobalava Z, Vida-Simiti L, Flather M, Shimokawa H, Ogawa H, Dellborg M, Rossi PRF, Troquay RPT, Libby P, Glynn RJ; CANTOS Trial Group. Antiinflammatory Therapy with Canakinumab for Atherosclerotic Disease. N Engl J Med. 2017 Sep 21;377(12):1119-1131. doi: 10.1056/NEJMoa1707914. Epub 2017 Aug 27. PMID 28845751
- [Background] Tardif JC, Kouz S, Waters DD, Bertrand OF, Diaz R, Maggioni AP, Pinto FJ, Ibrahim R, Gamra H, Kiwan GS, Berry C, Lopez-Sendon J, Ostadal P, Koenig W, Angoulvant D, Gregoire JC, Lavoie MA, Dube MP, Rhainds D, Provencher M, Blondeau L, Orfanos A, L'Allier PL, Guertin MC, Roubille F. Efficacy and Safety of Low-Dose Colchicine after Myocardial Infarction. N Engl J Med. 2019 Dec 26;381(26):2497-2505. doi: 10.1056/NEJMoa1912388. Epub 2019 Nov 16. PMID 31733140
- [Background] Nidorf SM, Fiolet ATL, Mosterd A, Eikelboom JW, Schut A, Opstal TSJ, The SHK, Xu XF, Ireland MA, Lenderink T, Latchem D, Hoogslag P, Jerzewski A, Nierop P, Whelan A, Hendriks R, Swart H, Schaap J, Kuijper AFM, van Hessen MWJ, Saklani P, Tan I, Thompson AG, Morton A, Judkins C, Bax WA, Dirksen M, Alings M, Hankey GJ, Budgeon CA, Tijssen JGP, Cornel JH, Thompson PL; LoDoCo2 Trial Investigators. Colchicine in Patients with Chronic Coronary Disease. N Engl J Med. 2020 Nov 5;383(19):1838-1847. doi: 10.1056/NEJMoa2021372. Epub 2020 Aug 31. PMID 32865380
- [Background] Tonino PA, De Bruyne B, Pijls NH, Siebert U, Ikeno F, van' t Veer M, Klauss V, Manoharan G, Engstrom T, Oldroyd KG, Ver Lee PN, MacCarthy PA, Fearon WF; FAME Study Investigators. Fractional flow reserve versus angiography for guiding percutaneous coronary intervention. N Engl J Med. 2009 Jan 15;360(3):213-24. doi: 10.1056/NEJMoa0807611. PMID 19144937
- [Background] Xu B, Tu S, Song L, Jin Z, Yu B, Fu G, Zhou Y, Wang J, Chen Y, Pu J, Chen L, Qu X, Yang J, Liu X, Guo L, Shen C, Zhang Y, Zhang Q, Pan H, Fu X, Liu J, Zhao Y, Escaned J, Wang Y, Fearon WF, Dou K, Kirtane AJ, Wu Y, Serruys PW, Yang W, Wijns W, Guan C, Leon MB, Qiao S, Stone GW; FAVOR III China study group. Angiographic quantitative flow ratio-guided coronary intervention (FAVOR III China): a multicentre, randomised, sham-controlled trial. Lancet. 2021 Dec 11;398(10317):2149-2159. doi: 10.1016/S0140-6736(21)02248-0. Epub 2021 Nov 4. PMID 34742368
- [Background] Huang AL, Maggiore PL, Brown RA, Turaga M, Reid AB, Merkur J, Blanke P, Leipsic JA. CT-Derived Fractional Flow Reserve (FFRCT): From Gatekeeping to Roadmapping. Can Assoc Radiol J. 2020 May;71(2):201-207. doi: 10.1177/0846537119893752. Epub 2020 Jan 24. PMID 32063007
- [Background] Tscharre M, Gremmel T. Antiplatelet Therapy in Coronary Artery Disease: Now and Then. Semin Thromb Hemost. 2023 Apr;49(3):255-271. doi: 10.1055/s-0042-1758821. Epub 2022 Dec 1. PMID 36455618
- [Background] Valgimigli M, Bueno H, Byrne RA, Collet JP, Costa F, Jeppsson A, Juni P, Kastrati A, Kolh P, Mauri L, Montalescot G, Neumann FJ, Petricevic M, Roffi M, Steg PG, Windecker S, Zamorano JL, Levine GN; ESC Scientific Document Group; ESC Committee for Practice Guidelines (CPG); ESC National Cardiac Societies. 2017 ESC focused update on dual antiplatelet therapy in coronary artery disease developed in collaboration with EACTS: The Task Force for dual antiplatelet therapy in coronary artery disease of the European Society of Cardiology (ESC) and of the European Association for Cardio-Thoracic Surgery (EACTS). Eur Heart J. 2018 Jan 14;39(3):213-260. doi: 10.1093/eurheartj/ehx419. No abstract available. PMID 28886622
- [Background] Krittanawong C, Johnson KW, Rosenson RS, Wang Z, Aydar M, Baber U, Min JK, Tang WHW, Halperin JL, Narayan SM. Deep learning for cardiovascular medicine: a practical primer. Eur Heart J. 2019 Jul 1;40(25):2058-2073. doi: 10.1093/eurheartj/ehz056. PMID 30815669
- [Background] Ambale-Venkatesh B, Yang X, Wu CO, Liu K, Hundley WG, McClelland R, Gomes AS, Folsom AR, Shea S, Guallar E, Bluemke DA, Lima JAC. Cardiovascular Event Prediction by Machine Learning: The Multi-Ethnic Study of Atherosclerosis. Circ Res. 2017 Oct 13;121(9):1092-1101. doi: 10.1161/CIRCRESAHA.117.311312. Epub 2017 Aug 9. PMID 28794054
- [Background] Pescatello LS, Wu Y, Panza GA, Zaleski A, Guidry M. Development of a Novel Clinical Decision Support System for Exercise Prescription Among Patients With Multiple Cardiovascular Disease Risk Factors. Mayo Clin Proc Innov Qual Outcomes. 2020 Oct 22;5(1):193-203. doi: 10.1016/j.mayocpiqo.2020.08.005. eCollection 2021 Feb. PMID 33718793
- [Background] Rosende A, DiPette DJ, Martinez R, Brettler JW, Rodriguez G, Zuniga E, Ordunez P. HEARTS in the Americas clinical pathway. Strengthening the decision support system to improve hypertension and cardiovascular disease risk management in primary care settings. Front Cardiovasc Med. 2023 Apr 26;10:1102482. doi: 10.3389/fcvm.2023.1102482. eCollection 2023. PMID 37180772